CLINICAL TRIAL: NCT02500498
Title: Safety Profile of Nulojix in Home Infusion Settings
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: BiologicTx, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IM103-370
Record Dates: First submitted 2015-07-15; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nulojix

SUMMARY:
The study is a retrospective cohort study that utilizes medical records from the BiologicTx. Data accrual starts upon initial home infusion nurse visit until the most recent home infusion nurse visit. Infusion related adverse events are quantified as number of patients with adverse event over the total number of patients and number of event over total number of home infusion visits.

ELIGIBILITY:
Inclusion Criteria:

* All adult kidney-only transplant recipients currently receiving NULOJIX in BiologicTx home infusion service settings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Home infusion service visit
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of infusion related serious adverse events in adult kidney-only transplant recipients who are treated with belatacept in home infusion settings | 24 hours after the date of a home infusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx